CLINICAL TRIAL: NCT03811275
Title: Functional Outcomes Following Task-based and VR Action Observation Interventions for Adults With Chronic Hemiparesis
Brief Title: Task or Virtual Reality Intervention for Improving UE Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped during the COVID-19 Pandemic in March 2020 to prevent transmission. It did not reopen due to aging of the virtual reality technology.
Sponsor: Idaho State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IdahoSU
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-05

CONDITIONS: Upper Extremity Paresis; Hemiplegia and/or Hemiparesis Following Stroke; Hemiplegic Cerebral Palsy
Keywords: upper extremity recovery of function; action observation; virtual reality; task-based intervention
MeSH Terms: conditions — Paresis | interventions — potassium channel subfamily K member 3

STUDY DESIGN:
Intervention Model Description: All participants will receive both interventions (A and B) and will be randomly assigned to the sequence in which they receive them (AB or BA).
Who Masked: Investigator
Masking Description: The occupational therapist providing all of the functional assessments will be blinded to sequence of interventions provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence #1 (Experimental): Participants will receive nine 30 minute sessions (over 3 weeks) of intervention A followed by nine 30 minute sessions (over 3 weeks) of intervention B.
  Interventions: Behavioral: Virtual Reality (A) then Task (B)
- Sequence #2 (Experimental): Participants will receive nine 30 minute sessions (over 3 weeks) of intervention B followed by nine 30 minute sessions (over 3 weeks) of intervention B.
  Interventions: Behavioral: Task (B) then Virtual Reality (A)

INTERVENTIONS:
Behavioral: Virtual Reality (A) then Task (B) — Participants will use their intact arm to perform virtual reality tasks while perceiving a reflected virtual image of their paretic arm.
  Arms: Sequence #1
Behavioral: Task (B) then Virtual Reality (A) — Participants will use their paretic arm to perform real tasks in a structured environment, with a practice and feedback schedule organized by a physical or occupational therapist, or graduate student.
  Arms: Sequence #2

SUMMARY:
People with one arm that does not function well due to a stroke, head injury, or cerebral palsy, and a fully functional other arm, will be randomly assigned to receive one of the two interventions first, followed by the other intervention. The two interventions include a task-based intervention and a virtual reality intervention that provides a reflected image of the involved arm. The task-based intervention will consist of setting up activities of interest to be done using the involved arm and structuring practice and meaningful feedback to assist learning. The virtual reality intervention will consist of the person wearing the virtual reality device and practicing virtual tasks using the intact arm while seeing the involved arm. Intervention sessions will last approximately 30 minutes and will be held 3 times/week for 3 weeks each for a total of 9 sessions for each intervention. Testing of the involved arm's function will be done before the interventions, after receiving 9 sessions of each intervention, and one month after completing the second intervention received.

DETAILED DESCRIPTION:
Potential participants will be screened for age, history of stroke, brain injury, or cerebral palsy, and having one functional arm and one poorly functioning arm by phone. Those who meet the basic criteria will be scheduled for an Intake Evaluation consisting of obtaining voluntary informed consent, complete a demographic survey, visual field testing, cognitive screening, perceptual testing, and an arm/hand function test. Participants who meet the inclusion criteria will be scheduled for a Preliminary Evaluation.

The Preliminary Evaluation will measure the current motor control ability, perception of level of disability, and amount of active and passive motion in the involved arm.

Participants will participate in the first form of intervention (randomly assigned) for three 30 minute sessions per week for 3 weeks (total of 9 sessions) and be re-evaluated using the same tests conducted during the Preliminary Evaluation with the addition of the arm/hand function test conducted during the initial screening.

Participants will participate in the second form of intervention for three 30 minute sessions per week for 3 weeks (total of 9 sessions) and be re-evaluated using the same tests conducted following the first intervention.

One month after completing the second form of intervention, participants will be re-evaluated using the same tests used following the second intervention and will also receive a semi-structured interview regarding their thoughts and experiences during the study and their perceptions of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 89 years old
* One arm not fully functional due to a stroke, brain injury, or cerebral palsy
* More than 1 year since neurologic even that impaired arm function

Exclusion Criteria:

* Cognitive impairment
* visual field loss (homonymous hemianopsia)
* perceptual deficits (MVPT4 lower than 2 standard deviations from the norm)
* Seizure disorder
* Currently receiving rehabilitation services (PT or OT) for the involved arm.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-08 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (UE portion) | 1st week, 4 weeks, 8 weeks, 12 weeks
  Performance-based measure of arm impairment post stroke; a positive change in score indicates improvement
Change in Box & Block Test | 1st week, 4 weeks, 8 weeks, 12 weeks
  Measures unilateral gross manual dexterity; a positive change in score indicates improvement
Change in Stroke Impact Scale 3.0 | 1st week, 4 weeks, 8 weeks, 12 weeks
  Self-report health status measure; The Total Score and Subscale Scores range from 0 - 100 with higher scores indicating less perceived impact of the stroke on function and participation (positive change in scores indicate improvement)

SECONDARY OUTCOMES:
Change in Active and Passive Range of Motion | 1st week, 4 weeks, 8 weeks, 12 weeks
  Goniometric measures of active and passive range of motion of the elbow extension, wrist extension, and thumb radial abduction.
Semi-structured interview | 12 weeks
  Qualitative measure of the participant's perception of change in arm function after participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Devine, PT, DPT, MS, Principal Investigator — Idaho State University
Locations (1):
- Nancy L Devine, Pocatello, Idaho, United States

IPD SHARING:
Plan to Share IPD: No